CLINICAL TRIAL: NCT02229565
Title: Molecular Mechanisms Underlying Prostate Cancer Disparities.
Acronym: GENCADE
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00053535
Record Dates: First submitted 2014-06-12; First posted 2014-09-01 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate biopsy; prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Biopsy; Prostatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Caucasian: Caucasian subjects having a biopsy or prostatectomy.
  Interventions: Device: Biopsy or prostatectomy
- African American: African American subjects having a biopsy or prostatectomy.
  Interventions: Device: Biopsy or prostatectomy

INTERVENTIONS:
Device: Biopsy or prostatectomy

SUMMARY:
The purpose of this study is to further elucidate the molecular mechanisms underlying prostate cancer disparities. In previous work the investigators have identified a set of differentially deregulated genes in African American versus Caucasian American prostate cancer. Based on these findings, they hypothesize that they will be able to validate these targets, originally identified in the previous work conducted at The George Washington University Medical Center, in an independent Duke University Medical Center cohort of prostate cancer specimens. In addition, the investigators hypothesize that they will be able to discover novel targets in the Duke University Medical Center cohort of prostate cancer specimens because of regional differences.

DETAILED DESCRIPTION:
Individual patient African American and Caucasian American prostate biopsy cores or surgical specimens will be obtained from the following procedures: transrectal ultrasound biopsy of the prostate (TRUSBxP), MR fusion biopsy, intra-operatively (IO) at the time of prostatectomy. Using cellular DNA and RNA, isolated from prostate cancer and patient-matched normal prostate biopsy cores or surgical specimens, the investigators will perform ancestral genotyping, exon arrays, targeted RNA sequencing, and epigenetic analyses. As controls, blood will also be collected. Genomic data from blood and tumor tissue will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Suspected malignancy of prostate cancer
* Self-reported race of African American or Caucasian American
* Age >/= 18 years
* Able to read, understand and sign an informed consent document

Exclusion Criteria:

* Collected tumor tissue is inadequate for DNA and RNA analysis and/or is not positive for adenocarcinoma of the prostate.
* Patients with prior systemic therapy will not be eligible for the study, i.e. radiation or chemo or immunotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes African American and Caucasian American patients (self-reported) undergoing clinically indicated diagnostic biopsies for a suspected prostate malignancy or intra-operative biopsies of patients undergoing clinically indicated prostatectomy for a confirmed prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Proportion of high and low expression of identified gene targets in Caucasian and African American specimens | up to 2 years
  Total RNA will be interrogated for mRNA expression patterns with the Affymetrix Human Exon 1.0 ST GeneChip. Microarray data will be normalized by quantile normalization with background correction. Targeted RNA sequencing of the previously identified genetic factors specific to African American prostate cancer will confirm altered expression and alternative splicing in these deregulated genes. The Agilent Technologies SureSelect RNA Custom Capture Kit will capture and sequence transcripts. Epigenetic analyses of the genetic factors specific to African American prostate cancer will identify DNA methylation and histone modification patterns in these deregulated genes. The Sequenom EpiTYPER will screen for differential methylation and methylation differences will be quantified using pyrosequencing. Differential histone modification patterns will be explored. Analysis will be performed on 33 prostate cancer biopsy specimens from each of 6 groups stratified by race and Gleason grade.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Patierno, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States